CLINICAL TRIAL: NCT05737394
Title: Laparoscopy-guided Versus Ultrasound-guided Transversus Abdominis Plane (TAP) Block in Pediatric Laparoscopy: a Randomized, Controlled Trial
Brief Title: Lap-guided vs Us-guided TAP Block in Pediatric Laparoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vittore Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Anna Camporesi, Principal Investigator, Vittore Buzzi Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/ST/264
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain
Keywords: tap block; laparoscopy; pediatric surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopy-guided TAP Block (Experimental): Patients will receive surgically-placed TAP block right after pneumoperitoneum induction and before Trocar insertion with levobupivacaine 0.25%, 0.5 ml/kg.
  Interventions: Procedure: Laparoscopic-guided TAP Block
- Ultrasound-guided TAP Block (Active Comparator): Patients will receive ultrasound-guided TAP block performed after anesthetic induction and before surgical incision with levobupivacaine 0.25%, 0.5 ml/kg.
  Interventions: Procedure: Ultrasound-guided TAP Block

INTERVENTIONS:
Procedure: Laparoscopic-guided TAP Block — Laparoscopically-assisted placement of block
  Arms: Laparoscopy-guided TAP Block
Procedure: Ultrasound-guided TAP Block — Ultrasound-assisted placement of block
  Arms: Ultrasound-guided TAP Block

SUMMARY:
Transversus Abdominis Plane (TAP) block is commonly used to control pain in laparoscopic procedures. It is usually administered with ultrasound guide but it can be also administered with laparoscopic assistance under direct visualization.

Aim of the present study is determining if the lap-assisted TAP is superior to the us-guided TAP Block in pain control in the immediate postoperative phase as well at 1 and 6 hours post surgery.

DETAILED DESCRIPTION:
Although pain in laparoscopic procedures has been demonstrated to be inferior to that of laparotomic ones, it is still produced because of rapid distension of peritoneum, visceral manipulation, irritation and traction of vessels and phrenic nerves, presence of residual gas and inflammatory mediators.

Analgesia can be achieved with multimodal techniques, which include oral or intravenous drugs as well as loco-regional anesthesia techniques.

The abdominal wall has three muscle layers: external and internal obliques, and transversus abdominis. They are innervated by mixed somatic nerves that course between the transversus abdominis and the internal oblique muscles.

Transversus Abdominis Plane Block is a regional analgesia technique which consists of injecting local anaesthetics between the transversus abdominis and internal oblique muscles, providing analgesia to the parietal peritoneum, skin and muscles of the anterior abdominal wall. It can provide benefit in both open and laparoscopic procedures and it is a safe technique, with a very low reported rate of complications.

Three major techniques are used to perform the Transversus Abdominis Plane (TAP) block-a landmark-based, an ultrasound-guided, and a surgical- placed TAP block.

Although the landmark technique is easy to perform, it might be complicated by inadvertent intraperitoneal organ damage.

Surgically administered Transversus Abdominis Plane (TAP) blocks have been performed by surgeons intraoperatively using the transperitoneal approach, accessing the Transversus Abdominis Plane (TAP) from the inside of the abdominal wall. Direct visualization of the needle and local anaesthetic spread may help to increase the accuracy as well as eliminating the risk of intraabdominal organ injury and is technically less difficult. It is however necessarily placed after incision and pneumoperitoneum establishment.

Ultrasound-guided Transversus Abdominis Plane (TAP) block on the other side can be performed prior to incision and pneumoperitoneum, thus avoiding nociception from the very beginning.

Aim of the present prospective, randomised, single center controlled study is to compare postoperative analgesic efficacy of laparo-assisted vs ultrasound-guided Transversus Abdominis Plane (TAP) block in pediatric laparoscopic procedures. Primary outcome will be the comparison of pain scores between groups upon arrival to Post-Anesthesia Care Unit (PACU).

Secondary outcomes are:

* pain scores at 1 and 6 hours after surgery
* general anesthesia requirements, as defined by Minimum Alveolar Concentration-hour (MAC_hour)
* intraoperative opiod consumption
* complication rates
* time to block completion

ELIGIBILITY:
Inclusion Criteria:

* Age<= 18 yrs
* Elective or urgent laparoscopic surgical procedures including hernia repair, appendectomy, cholecystectomy, piloromyotomy, Nissen fundoplication, varicocelectomy
* ASA Status I and II

Exclusion Criteria:

* absence of parental consent
* ASA Status III-VI
* Presence of neurological disability affecting spontaneous mobility
* Previous surgical procedures on the abdominal wall (e.g. gastroschisis repair)
* Foreseen surgical duration bigger than 4 hours
* Conversion to laparotomy
* Use of concomitant other regional anesthesia technique (e.g. neuraxial or peripheral)

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-28 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain scores in PACU | Post-Anesthesia Care Unit - immediately after end of surgery
  Pain will be measured with FLACC scale (0-10 points; 0 no pain, 10 maximal pain) by operators blinded to the TAP technique

SECONDARY OUTCOMES:
Pain scores at 1 and 6 hours post-op | first 6 hours post - op
  Comparison of pain scores measured with FLACC scale (0-10 points; 0 no pain, 10 maximal pain)by operators blinded to the TAP technique
Intraoperative opioids requirements | Intraoperative
  Comparison of need for additional boluses of intraoperative opioids if HR raises more than 10% of baseline
General anesthetic requirements | Intraoperative
  Comparison of MAC-hour in the two groups
Time to Block completion | Intraoperative
  Comparison of time needed to place the block between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Vittore Buzzi Children's Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No